CLINICAL TRIAL: NCT00900731
Title: A 12-week Treatment, Multicenter, Randomized, Parallel-group, Blinded, Double-dummy Study to Compare the Efficacy and Safety of Indacaterol (150 µg Once Daily [od]) Delivered Via a Single Dose Dry Powder Inhaler (SDDPI) With Tiotropium (18 µg od) Delivered Via a HandiHaler®, in Patients With Moderate-to-severe COPD
Brief Title: A Study to Compare the Lung Effect of Indacaterol and Tiotropium in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: INTENSITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149B2350
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; indacaterol; beta 2 agonist; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Indacaterol 150 µg (Experimental): Participants received indacaterol 150 μg delivered via a single-dose dry-powder inhaler (SDDPI) plus placebo to tiotropium delivered via the manufacturer's proprietary inhalation device (HandiHaler®) once daily in the morning. Participants were permitted to take salbutamol/albuterol as a rescue medication.
  Interventions: Drug: Indacaterol 150 μg; Drug: Placebo to tiotropium
- Tiotropium 18 µg (Active Comparator): Participants received tiotropium 18 μg delivered via the manufacturer's proprietary inhalation device (HandiHaler®) plus placebo to indacaterol delivered via a single-dose dry-powder inhaler (SDDPI) once daily in the morning. Participants were permitted to take salbutamol/albuterol as a rescue medication.
  Interventions: Drug: Tiotropium 18 μg; Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol 150 μg — Indacaterol 150 μg was provided in powder filled capsules with a single dose dry powder inhaler (SDDPI).
  Arms: Indacaterol 150 µg
Drug: Tiotropium 18 μg — Tiotropium 18 μg was provided in powder filled capsules with the manufacturer's proprietary inhalation device (HandiHaler®).
  Arms: Tiotropium 18 µg
Drug: Placebo to indacaterol — Placebo to indacaterol was provided in powder filled capsules with a single dose dry powder inhaler (SDDPI).
  Arms: Tiotropium 18 µg
Drug: Placebo to tiotropium — Placebo to tiotropium was provided in powder filled capsules with the manufacturer's proprietary inhalation device (HandiHaler®).
  Arms: Indacaterol 150 µg

SUMMARY:
This study compared the lung effects of indacaterol to those of tiotropium in patients with moderate to severe chronic obstructive pulmonary disease (COPD) over a 12 week period.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of COPD (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2007) and:

* a) Smoking history of at least 10 pack-years
* b) Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥ 30% of the predicted normal value
* c) Post-bronchodilator FEV1/FVC (forced vital capacity) < 70%

Exclusion Criteria:

* Patients who have received systemic corticosteroids or antibiotics and/or was hospitalized for a COPD exacerbation in the 6 weeks prior to screening
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1598 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (212):
- United States (25):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigator Site, Jasper, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigator Site, Anaheim, California
  - Novartis Investigator Site, Stockton, California
  - Novartis Investigator Site, Walnut Creek, California
  - Novartis Investigator Site, Fort Collins, Colorado
  - Novartis Investigator Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigator Site, Normal, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Center, Saint Charles, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Larchmont, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Richmond, Virginia
- Austria (3):
  - Novartis Investigator Site, Feldbach
  - Novartis Investigator Site, Gänserndorf
  - Novartis Investigator Site, Hallein
- Belgium (9):
  - Novartis Investigator Site, Brussels
  - Novartis Investigator Site, Gilly
  - Novartis Investigator Site, Jambes
  - Novartis Investigator Site, Jette
  - Novartis Investigator Site, Liège
  - Novartis Investigator Site, Montigny-le-Tilleul
  - Novartis Investigator Site, Ostend
  - Novartis Investigator Site, Sankt Vith
  - Novartis Investigator Site, Yvoir
- Canada (7):
  - Novartis Investigator Site, Calgary
  - Novartis Investigative Site, Greater Sudbury
  - Novartis Investigative Site, Mississauga
  - Novartis Investigative Site, Moncton
  - Novartis Investigative Site, New Market
  - Novartis Investigative SIte, Québec
  - Novartis Investigative Site, Saint Romuald
- Colombia (3):
  - Novartis Investigator Site, Barranquilla
  - Novartis Investigator Site, Bogotá
  - Novartis Investigator Site, Medellín
- Denmark (7):
  - Novartis Investigator Site, Aalborg
  - Novartis Investigator Site, Frederiksberg
  - Novartis Investigator Site, Næstved
  - Novartis Investigator Site, Roskilde
  - Novartis Investigator Site, Sønderborg
  - Novartis Investigator Site, Viborg
  - Novartis Investigator Site, Værløse
- Finland (6):
  - Novartis Investigator Site, Helsinki
  - Novartis Investigator Site, Jyväskylä
  - Novartis Investigator Site, Lahti
  - Novartis Investigator Site, OYS
  - Novartis Investigator Site, Pori
  - Novartis Investigator Site, Turku
- France (14):
  - Novartis Investigative Site, Ambroise
  - Novartis Investigative Site, Antibes
  - Novartis Investigator Site, Beuvry
  - Novartis Investigator Site, Ferolles-Attily
  - Novartis Investigative Site, Montpellier
  - Novartis Investigator Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigator Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigator Site, Pierre-Bénite
  - Novartis Investigative Site, Suresnes
  - Novartis Investigator Site, Vandoeuvre Les Nancys
- Germany (35):
  - Novartis Investigator Site, Bergisch Gladbach
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Bochum
  - Novartis Investigator Site, Bonn
  - Novartis Investigator Site, Buchholz
  - Novartis Investigator Site, Coburg
  - Novartis Investigator Site, Düren
  - Novartis Investigator Site, Eggenfelden
  - Novartis Investigator Site, Eschwege
  - Novartis Investigator Site, Euskirchen
  - Novartis Investigator Site, Freudenberg
  - Novartis Investigator Site, Fürth
  - Novartis Investigator Site, Gelsenkirchen
  - Novartis Investigator Site, Gummersbach
  - Novartis Investigator Site, Hagen
  - Novartis Investigator Site, Halle
  - Novartis Investigator Site, Hamburg
  - Novartis Investigator Site, Hanover
  - Novartis Investigator Site, Hoyerswerda
  - Novartis Investigator Site, Kassel
  - Novartis Investigative Site, Landsberg
  - Novartis Investigator Site, Leipzig
  - Novartis Investigator Site, Mainz
  - Novartis Investigator Site, Munich
  - Novartis Investigator Site, Oranienburg
  - Novartis Investigator Site, Radebeul
  - Novartis Investigator Site, Ratingen
  - Novartis Investigator Site, Ruhmannsfelden
  - Novartis Investigator Site, Rüsselsheim am Main
  - Novartis Investigator Site, Solingen
  - Novartis Investigator Site, Stockach
  - Novartis Investigator Site, Teterow
  - Novartis Investigator Site, Vilshofen
  - Novartis Investigator Site, Wallerfing
  - Novartis Investigator Site, Wissen
- Novartis Investigator Site, Athens, Greece
- Hungary (6):
  - Novartis Investigative Site, Budapest
  - Novartis Investigator Site, Budapest
  - Novartis Investigator Site, Debrecen
  - Novartis Investigative Site, Farkasgyepű
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigator Site, Szolnok
- Israel (2):
  - Novartis Investigator Site, Haifa
  - Novartis Investigator Site, Petah Tikva
- Italy (8):
  - Novartis Investigator Site, Ancona
  - Novartis Investigator Site, Foggia
  - Novartis Investigative Site, Milan
  - Novartis Investigator Site, Milan
  - Novartis Investigative Site, Pavia
  - Novartis Investigator Site, Pavia
  - Novartis Investigative Site, Pisa
  - Novartis Investigator Site, Pisa
- Mexico (3):
  - Novartis Investigative Site, Huxquilucan
  - Novartis Investigator Site, Mexico City
  - Novartis Investigative Site, San Luis Potosí City
- Norway (15):
  - Novartis Investigative Site, Ålesund
  - Novartis Investigator Site, Ålesund
  - Novartis Investigator Site, Drammen
  - Novartis Investigator Site, Follebu
  - Novartis Investigative Site, Kongsberg
  - Novartis Investigator Site, Kongsberg
  - Novartis Investigator Site, Kongsvinger
  - Novartis Investigator Site, Lierskogen
  - Novartis Investigative Site, Oslo
  - Novartis Investigator Site, Oslo
  - Novartis Investigator Site, Sandvika
  - Novartis Investigative Site, Skedsmokorset
  - Novartis Investigator Site, Stavanger
  - Novartis Investigative Site, Trondheim
  - Novartis Investigator Site, Trondheim
- Poland (7):
  - Novartis Investigator Site, Gdansk
  - Novartis Investigator Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigator Site, Krakow
  - Novartis Investigator Site, Piekary Śląskie
  - Novartis Investigator Site, Warsaw
  - Novartis Investigator Site, Wroclaw
- Russia (9):
  - Novartis Investigator Site, Barnaul
  - Novartis Investigator Site, Kazan'
  - Novartis Investigator Site, Novosibirsk
  - Novartis Investigator Site, Petrozavodsk
  - Novartis Investigator Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigator Site, Saint Petersburg
  - Novartis Investigator Site, Samara
  - Novartis Investigator Site, Yekaterinburg
- Slovakia (7):
  - Novartis Investigator Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigator Site, Košice
  - Novartis Investigator Site, Kráľovský Chlmec
  - Novartis Investigator Site, Nitra
  - Novartis Investigative Site, Prešov
  - Novartis Investigator Site, Zvolen
- Spain (19):
  - Novartis Investigative Site, Alcorcón
  - Novartis Investigator Site, Alicante
  - Novartis Investigator Site, Badalona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Begonte
  - Novartis Investigator Site, Burgos
  - Novartis Investigator Site, Canet de Mar
  - Novartis Investigator Site, Cáceres
  - Novartis Investigator Site, el Prat de Llobregat
  - Novartis Investigative Site, Fuenlabrada
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Madrid
  - Novartis Investigator Site, Mataró
  - Novartis Investigator Site, Plasencia
  - Novartis Investigative Site, Ponferrada
  - Novartis Investigative Site, Pontevedra
  - Novartis Investigative Site, Santander
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Vila-real
- Switzerland (5):
  - Novartis Investigator Site, Basel
  - Novartis Investigator Site, Bellinzona
  - Novartis Investigator Site, Lugano
  - Novartis Investigator Site, Muenchenstein
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (11):
  - Novartis Investigator Site, Altunizade
  - Novartis Investigator Site, Ankara
  - Novartis Investigative Site, Aydin
  - Novartis Investigator Site, Büyükçekmece / Ýstanbul
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigator Site, Istanbul
  - Novartis Investigator Site, Kahramanmaraş
  - Novartis Investigative Site, Mecidiyekoy/Istanbul
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Soke / Aydin
  - Novartis Investigative Site, Yenisehir/Izmir
- United Kingdom (10):
  - Novartis Investigator Site, Ash Vale
  - Novartis Investigator Site, Ashford
  - Novartis Investigator Site, Bolton
  - Novartis Investigator Site, Boscastle
  - Novartis Investigator Site, Bradford
  - Novartis Investigator Site, Chertsey
  - Novartis Investigator Site, East Horsley
  - Novartis Investigator Site, Newcastle upon Tyne
  - Novartis Investigator Site, Plymouth
  - Novartis Investigator Site, Watford

REFERENCES:
- [Derived] Buhl R, Dunn LJ, Disdier C, Lassen C, Amos C, Henley M, Kramer B; INTENSITY study investigators. Blinded 12-week comparison of once-daily indacaterol and tiotropium in COPD. Eur Respir J. 2011 Oct;38(4):797-803. doi: 10.1183/09031936.00191810. Epub 2011 May 26. PMID 21622587

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1598 participants were randomized. 3 participants in the Indacaterol group and 2 participants in the Tiotropium group did not receive study medication.
Period: Overall Study
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg
Started | 797 (Randomized participants) | 801
Safety Set: Received Study Drug | 794 | 799
Completed | 737 | 740
Not Completed | 60 | 61
Not completed — Adverse Event | 31 | 27
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Protocol Deviation | 8 | 11
Not completed — Administrative Problems | 5 | 4
Not completed — Abnormal Test Procedure Result(s) | 3 | 0
Not completed — Abnormal Laboratory Value(s) | 2 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Lack of Efficacy | 1 | 3
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg | Total
Number analyzed (Participants) | 794 | 799 | 1593
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline Measures used the safety population that consisted of all participants who received at least one dose of study drug.
  years | 63.6 (8.60) | 63.4 (8.29) | 63.5 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 261 | 500
  Male | 555 | 538 | 1093

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at End of Treatment (Week 12)
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 was defined as the average of the 23 hour 10 minute and 23 hour 45 minute post-dose FEV1 readings. Mixed model used baseline FEV1, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, FEV1 prior to and 1 hour post inhalation of ipratropium, and inhaled corticosteroid use at baseline as covariates.
Time Frame: End of treatment (Week 12)
Population: Per-protocol population included all participants who received at least one dose of study medication without any major protocol deviations. The endpoint was analyzed only for those participants who had data for this outcome measure. Missing data were imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg
Number analyzed (Participants) | 562 | 595
Liters | 1.44 (0.010) | 1.43 (0.010)

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Time) Area Under the Curve (AUC) From 5 Minutes to 4 Hours Post-dose at the End of Treatment (Week 12)
Description: Spirometry was conducted according to internationally accepted standards. FEV1 was measured at 5 and 30 minutes; and 1, 2, and 4 hours post-dose on Week 12. Standardized FEV1 AUC (5 minutes-4 hour) post-dose at week 12 was calculated based on the trapezoidal rule, and was adjusted for the area per time unit by using the scheduled time of measurements for FEV1. Mixed model used baseline FEV1, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, FEV1 prior to and 1 hour post inhalation of ipratropium, and inhaled corticosteroid use at baseline as covariates.
Time Frame: 5 minutes to 4 hours post-dose at the end of treatment (week 12)
Population: Full analysis set included all participants who received at least one dose of study medication. The endpoint was analyzed only for those participants who had data at week 12 for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg
Number analyzed (Participants) | 685 | 692
Liter | 1.51 (0.010) | 1.52 (0.010)

3. Secondary Outcome: Transition Dyspnea Index (TDI) Focal Score After 12 Weeks of Treatment
Description: TDI focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort. Each domain is scored from -3 (major deterioration) to 3 (major improvement) to give an overall TDI focal score of -9 to 9 with a negative score indicating a deterioration from baseline. A 1 unit difference in the TDI focal score is clinically significant. Mixed model used baseline dyspnea index, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, FEV1 prior to and 1 hour post inhalation of ipratropium, and inhaled corticosteroid use at baseline as covariates.
Time Frame: 12 weeks
Population: Full Analysis Set included all randomized participants who received at least one dose of study drug. The endpoint was analyzed only for those participants who had data at week 12 for this outcome measure. Missing data were imputed using Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg
Number analyzed (Participants) | 729 | 737
Score on a scale | 2.01 (0.178) | 1.43 (0.178)

4. Secondary Outcome: Quality of Life Assessment With St. George's Respiratory Questionnaire (SGRQ) Total Score After 12 Weeks of Treatment
Description: SGRQ is a health related quality of life questionnaire consisting of 50 items in three domains: symptoms (frequency and severity), activity (that cause or are limited by breathlessness) and impacts (social functioning & psychological disturbances resulting from airway disease). The total score is 0 to 100 with a higher score indicating greater impairment of health status. Mixed model used baseline SGRQ, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, FEV1 prior to and 1 hour post inhalation of ipratropium, and inhaled corticosteroid use at baseline as covariates.
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg
Number analyzed (Participants) | 743 | 753
Score on a scale | 37.1 (0.56) | 39.2 (0.55)

5. Secondary Outcome: Change From Baseline in the Mean Number of Puffs Per Day of Rescue Medication Over the Study Duration (From Day 1 to Week 12)
Description: Participants recorded the number of puffs of rescue medication taken in the previous 12 hours each morning and evening in an electronic diary. The number of puffs per day over the 12 weeks of treatment was divided by the number of days to derive the mean number per day of puffs of rescue medication for each participant. Mixed model used baseline number of puffs per day of rescue medication, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, FEV1 prior to and 1 hour post inhalation of ipratropium, and inhaled corticosteroid use at baseline as covariates.
Time Frame: Baseline, up to 12 weeks
Population: Full analysis set included all participants who received at least 1 dose of study medication. The endpoint was analyzed only for those participants who had data at baseline and at week 12 for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg
Number analyzed (Participants) | 740 | 747
Puffs | -1.40 (0.097) | -0.85 (0.097)

6. Secondary Outcome: Change From Baseline in the Mean Number Per Day of Daytime Puffs of Rescue Medication Over the Study Duration (From Day 1 to Week 12)
Description: Participants recorded the number of puffs of rescue medication taken in the previous 12 hours each evening in an electronic diary. The number of daytime puffs per day over the 12 weeks of treatment was divided by the number of days to derive the mean number per day of daytime puffs of rescue medication for each participant. Mixed model used baseline number of daytime puffs per day of rescue medication, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, FEV1 prior to and 1 hour post inhalation of ipratropium, and inhaled corticosteroid use at baseline as covariates.
Time Frame: Baseline, up to 12 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg
Number analyzed (Participants) | 722 | 732
Puffs | -0.90 (0.063) | -0.59 (0.063)

7. Secondary Outcome: Change From Baseline in the Mean Number Per Day of Nighttime Puffs of Rescue Medication Over the Study Duration (From Day 1 to Week 12)
Description: Participants recorded the number of puffs of rescue medication taken in the previous 12 hours each morning in an electronic diary. The number of nighttime puffs per day over the 12 weeks of treatment was divided by the number of days to derive the mean number per day of nighttime puffs of rescue medication for each participant. Mixed model used baseline number of nighttime puffs per day of rescue medication, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, FEV1 prior to and 1 hour post inhalation of ipratropium, and inhaled corticosteroid use at baseline as covariates.
Time Frame: Baseline, up to 12 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg
Number analyzed (Participants) | 729 | 742
Puffs | -0.52 (0.043) | -0.28 (0.042)

8. Secondary Outcome: Percentage of Days With no Rescue Medication Use During the 12 Weeks of Treatment
Description: A day with no rescue medication was defined as any day in the diary that the participant used no puffs of rescue medication. The percentage of days with no rescue medication was calculated by dividing the number of days with no rescue medication over the 12 week treatment period by the number of evaluable days and multiplying by 100. Mixed model used baseline percentage of days with no rescue medication, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, FEV1 prior to and 1 hour post inhalation of ipratropium, and inhaled corticosteroid use at baseline as covariates.
Time Frame: Up to 12 weeks
Population: Full analysis set included all participants who received at least one dose of study medication. The endpoint was analyzed only for those participants who had data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | Indacaterol 150 µg | Tiotropium 18 µg
Number analyzed (Participants) | 725 | 738
Percentage of days | 46.1 (1.65) | 41.4 (1.64)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety set consisting of all participants who received at least one dose of study drug.
Groups:
- Indacaterol 150 μg: Participants received indacaterol 150 μg delivered via a single-dose dry-powder inhaler (SDDPI) plus placebo to tiotropium delivered via the manufacturer's proprietary inhalation device (HandiHaler®) once daily in the morning. Participants were permitted to take salbutamol/albuterol as a rescue medication.
- Tiotropium 18 μg: Participants received tiotropium 18 μg delivered via the manufacturer's proprietary inhalation device (HandiHaler®) plus placebo to indacaterol delivered via a single-dose dry-powder inhaler (SDDPI) once daily in the morning. Participants were permitted to take salbutamol/albuterol as a rescue medication.
Arm/Group | Indacaterol 150 μg | Tiotropium 18 μg
Serious Adverse Events (participants affected / at risk) | 22/794 | 30/799
Other Adverse Events (participants affected / at risk) | 80/794 | 61/799
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=794) | Tiotropium 18 μg (N=799)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Diabetic eye disease (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Vagus nerve paralysis (Nervous system disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=794) | Tiotropium 18 μg (N=799)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 80 | 61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.